CLINICAL TRIAL: NCT07369531
Title: The Impact of Two-Stage Turnbull-Cutait Pull-Through Coloanal Anastomosis on Stoma-free Survival in Low Rectal Anal-preserving Surgery: A Multicenter Randomized Controlled Trial (RC09-FIAS)
Brief Title: The Impact of Two-Stage Turnbull-Cutait Pull-Through Coloanal Anastomosis on Stoma-free Survival in Low Rectal Anal-preserving Surgery
Acronym: RC09-FIAS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Quan Wang, Principal Investigator (PI), The First Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC09-FIAS
Record Dates: First submitted 2025-12-28; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Rectal Cancer; Surgical Anastomosis; Survival , Tumor; Anal Function; Stoma
Keywords: Turnbull-Cutait anastomosis; Rectal neoplasms; Low anterior resection; Stoma-free survival
MeSH Terms: conditions — Rectal Neoplasms; Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LAR group (Active Comparator): First Surgery
  1. The inferior mesenteric artery is transected at its root.
  2. After mobilization to the levator ani hiatus, surgeons may choose to transect the intestinal tract using a linear cutting stapler under laparoscopy according to the location of the tumor's lower margin. Subsequently, a circular stapler is inserted transanally to perform sigmoid-colorectal anastomosis or sigmoid-anal canal anastomosis.
  3. If the tumor is adjacent to the anal canal, an intersphincteric resection (ISR) is required, and hand-sewn end-to-end sigmoid-anal canal anastomosis is completed transanally.
  4. All patients in the LAR group undergo a protective stoma, which is placed in the right lower quadrant through the rectus abdominis muscle as a loop ileostomy.
  Second Surgery The stoma reversal surgery for patients in the LAR group should be completed 3 to 4 months after the first surgery.
  Interventions: Procedure: LAR
- TCA group (Experimental): First Surgery
  1. Abdominal procedure: The inferior mesenteric artery is ligated at its root. The splenic flexure of the colon is mobilized.
  2. After mobilization to the levator ani hiatus and entry into the intersphincteric space, the procedure switches to transanal operation. The full thickness of the rectal wall is incised 1 cm above the lower edge of the tumor.
  5. The rectal tumor and sigmoid colon are pulled out transanally. The sigmoid colon is transected approximately 8 cm above the tumor to complete tumor resection. The distal sigmoid colon is pulled out 4-5 cm through the anus, and the four pre-placed marking sutures are secured to fix sigmoid colon to the anal canal stump.
  Second Surgery
  1. The second surgery for resecting the pulled-out intestinal segment is performed 7-11 days after the first operation. The pulled-out intestinal segment is transected approximately 2 mm caudal to the anal canal stump plane. Subsequently, end-to-end anastomosis is completed.
  Interventions: Procedure: Turnbull-Cutait anastomosis

INTERVENTIONS:
Procedure: Turnbull-Cutait anastomosis — First Surgery 1. Abdominal procedure: The inferior mesenteric artery is ligated at its root. The splenic flexure of the colon is mobilized. 2. After mobilization to the levator ani hiatus and entry into the intersphincteric space, the procedure switches to transanal operation. The full thickness of the rectal wall is incised 1 cm above the lower edge of the tumor. 5. The rectal tumor and sigmoid colon are pulled out transanally. The sigmoid colon is transected approximately 8 cm above the tumor to complete tumor resection. The distal sigmoid colon is pulled out 4-5 cm through the anus, and the four pre-placed marking sutures are secured to fix sigmoid colon to the anal canal stump. Second Surgery 1. The second surgery for resecting the pulled-out intestinal segment is performed 7-11 days after the first operation. The pulled-out intestinal segment is transected approximately 2 mm caudal to the anal canal stump plane. Subsequently, end-to-end anastomosis is completed.
  Other Names: TCA
  Arms: TCA group
Procedure: LAR — First Surgery 1. The inferior mesenteric artery is transected at its root. 2. After mobilization to the levator ani hiatus, surgeons may choose to transect the intestinal tract using a linear cutting stapler under laparoscopy according to the location of the tumor's lower margin. Subsequently, a circular stapler is inserted transanally to perform sigmoid-colorectal anastomosis or sigmoid-anal canal anastomosis. 3. If the tumor is adjacent to the anal canal, an intersphincteric resection (ISR) is required, and hand-sewn end-to-end sigmoid-anal canal anastomosis is completed transanally. 4. All patients in the LAR group undergo a protective stoma, which is placed in the right lower quadrant through the rectus abdominis muscle as a loop ileostomy.
  Second Surgery The stoma reversal surgery for patients in the LAR group should be completed 3 to 4 months after the first surgery.
  Arms: LAR group

SUMMARY:
The goal of this clinical trial is to explore the difference in 3-year stoma-free survival between the Turnbull-Cutait delayed coloanal anastomosis (TCA) surgery and the low anterior resection combined with protective stoma (LAR) surgery in patients with low rectal cancer, as well as the differences in anal function, surgical complications, and survival outcomes within 1 year after surgery. The main questions it aims to answer are:

1. Is TCA surgery superior to LAR surgery in improving the 3-year stoma-free survival of patients with low rectal cancer?
2. Are there differences in postoperative anal function (assessed by LARS score and Wexner score), quality of life (assessed by EORTC QLQ-CR29 questionnaire), surgical complications, pathological outcomes, and long-term survival (disease-free survival, time to recurrence, overall survival) between the two surgical methods? Researchers will compare the TCA group and the LAR group to see if TCA surgery can reduce the permanent stoma rate, improve postoperative anal function and quality of life, and ensure surgical safety and favorable tumor-related outcomes compared with LAR surgery.

Participants will:

1. Be randomly assigned to either the TCA group or the LAR group in a 1:1 ratio.
2. Receive the corresponding surgical intervention.
3. Complete regular follow-ups at 1 month, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 30 months, and 36 after the first surgery.
4. Provide relevant clinical data (perioperative, pathological, follow-up) as required.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with rectal cancer aged 18-75 years confirmed by pathological biopsy as adenocarcinoma;
2. Preoperative abdominal contrast-enhanced CT and pulmonary CT (or PET-CT) showed no evidence of distant metastasis;
3. Preoperative rectal MRI evaluation demonstrated that the tumor was located within 5cm below the anal margin, above the intermuscular groove between the internal and external anal sphincters (anal white line) by 1 cm, and without invasion of the external anal sphincter;
4. For tumors located above the levator ani hiatus, MRI evaluation showed cT1-3, cN0-1, M0, MRF (-); for tumors located below the levator ani hiatus, MRI evaluation showed cT1-2, cN0-1, M0, MRF (-). For patients who received neoadjuvant therapy, tumors above the levator ani hiatus were downstaged to ycT3NxM0 or below, and tumors below the levator ani hiatus were downstaged to ycT2NxM0 or below;
5. Patients underwent radical laparoscopic/robot-assisted total mesorectal excision (TME) or transanal total mesorectal excision (TaTME).

Exclusion Criteria:

1. Patients diagnosed with concurrent primary malignant tumors in any other organ or multiple distant colorectal cancers;
2. History of previous open surgery (non-minimally invasive procedures);
3. Failure to undergo preoperative rectal MRI evaluation and chest/abdominal imaging assessment, resulting in incomplete clinical staging of the tumor;
4. Pregnant patients or those with concurrent inflammatory bowel disease;
5. Preoperative patients with complete intestinal obstruction or requiring emergency surgery;
6. Preoperative evaluation necessitating combined organ resection;
7. Recent treatment for other malignancies;
8. Low rectal cancer classified as type IV in the Bordeaux classification system;
9. Preoperative pathological types of signet ring cell carcinoma, mucinous adenocarcinoma, anaplastic carcinoma, or poorly differentiated carcinoma.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
3-year stoma-free survival postoperatively | 3 years
  During the follow-up period, death from any cause or an irreducible enterostomy (whichever occurs first) was recorded. An irreducible enterostomy was defined as an event where the enterostomy had not been reduced by the end of the 3-year follow-up period, or at the time of loss to follow-up, or at the time of death.

SECONDARY OUTCOMES:
LARS grading | 3 months, 6 months, 9 months, 1 year, 2 years, 3 years
  The full name of LARS grading is Low Anterior Resection Syndrome grading, with its core assessment tool being the LARS score (Low Anterior Resection Syndrome score). This grading system categorizes patients into three levels based on the LARS score: no LARS (0-20 points), mild LARS (21-29 points), and severe LARS (30-42 points). It quantifies the severity of intestinal dysfunction following low anterior resection of the rectum, with higher scores indicating more severe dysfunction.
Wexner scale | 3 months, 6 months, 9 months, 1 year, 2 years, 3 years
  The Wexner scale, formally known as the Wexner Fecal Incontinence Rating Scale, is a commonly used tool for quantitatively assessing the severity of anal incontinence. The scoring range is 0-20 points, with 0 indicating normal and 20 indicating complete incontinence. Higher scores indicate more severe incontinence.
Quality of Life Questionnaire (EORTC QLQ-CR29) | 1 month, 6 months, 1 year
  The EORTC QLQ-CR29, formally known as the European Organization for Research and Treatment of Cancer Colorectal Cancer-Specific Quality of Life Questionnaire 29 Items, is used to assess health-related quality of life in colorectal cancer patients. The functional dimension score ranges from 0 to 100, with higher scores indicating better functional status. The symptom dimension score also ranges from 0 to 100, with higher scores indicating more severe symptoms.

OTHER OUTCOMES:
Types and Classification of Postoperative Complications | 3 years
  Both surgical complications should be recorded separately, with documentation including the type and severity of complications. Types include infection (incisional infection, pulmonary infection, urinary tract infection, etc.), hemorrhage, organ dysfunction (e.g., cardiac insufficiency, respiratory failure, renal impairment, etc.), anastomotic leakage, thrombosis (deep vein thrombosis, pulmonary embolism, etc.), gastrointestinal dysfunction (e.g., intestinal obstruction, diarrhea, constipation, etc.), and other adverse events directly or indirectly related to the surgery. The severity of complications is typically assessed using the Clavien-Dindo classification system.
Surgical duration | From the start of the procedure (e.g., skin incision) to the completion of the surgery (e.g., suturing the incision)
  The duration from the start of the procedure (e.g., skin incision) to the end of the procedure (e.g., completion of suture closure) is recorded in minutes.
Postoperative hospitalization duration | Perioperative
  The postoperative hospitalization duration for both procedures shall be recorded separately. The number of days a patient is hospitalized after surgery is calculated from the end of the procedure until discharge.
Hospitalization expenses | Perioperative
  The hospitalization costs for both surgical procedures shall be recorded separately. All medical expenses incurred during the patient's hospitalization period (including the surgical and postoperative recovery phases) shall be documented, covering surgical fees, anesthesia fees, medication fees, examination and testing fees (such as laboratory tests, imaging examinations, etc.), nursing fees, bed fees, medical device usage fees (such as implants, disposable consumables, etc.), and other treatment-related expenses.
Three-year disease-free survival after surgery | 3 years
  The observation window was defined as the period from the randomization date to the time of tumor recurrence in the patient, or death from any cause (whichever occurred first), or the last confirmed date of no recurrence and no death (censored date), with a follow-up period of 3 years after randomization.
Recurrence rate at 3 years postoperatively | 3 years
  The endpoint event was tumor recurrence in patients or death due to tumor recurrence. It refers to the time from the randomization date until the occurrence of tumor recurrence or death caused by tumor recurrence. Lost to follow-up during the follow-up period and deaths due to non-tumor recurrence causes were treated as censored values.
Three-year overall survival after surgery | 3 years
  The endpoint event was patient death from any cause. The time from the randomization date to patient death from any cause was calculated. Lost-to-follow-up during follow-up was treated as censored.

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Yamada K, Ogata S, Saiki Y, Fukunaga M, Tsuji Y, Takano M. Functional results of intersphincteric resection for low rectal cancer. Br J Surg. 2007;94(10):1272-7.
- [Background] Cohen R, Vernerey D, Bellera C, Meurisse A, Henriques J, Paoletti X, et al. Guidelines for time-to-event end-point definitions in adjuvant randomised trials for patients with localised colon cancer: Results of the DATECAN initiative. Eur J Cancer. 2020;130:63-71.
- [Background] David GG, Slavin JP, Willmott S, Corless DJ, Khan AU, Selvasekar CR. Loop ileostomy following anterior resection: is it really temporary? Colorectal Dis. 2010;12(5):428-32.
- [Background] Lindgren R, Hallböök O, Rutegård J, Sjödahl R, Matthiessen P. What is the risk for a permanent stoma after low anterior resection of the rectum for cancer? A six-year follow-up of a multicenter trial. Dis Colon Rectum. 2011;54(1):41-7.
- [Background] Bailey CM, Wheeler JM, Birks M, Farouk R. The incidence and causes of permanent stoma after anterior resection. Colorectal Dis. 2003;5(4):331-4.
- [Background] den Dulk M, Smit M, Peeters KC, Kranenbarg EM, Rutten HJ, Wiggers T, et al. A multivariate analysis of limiting factors for stoma reversal in patients with rectal cancer entered into the total mesorectal excision (TME) trial: a retrospective study. Lancet Oncol. 2007;8(4):297-303.
- [Background] Dinnewitzer A, Jäger T, Nawara C, Buchner S, Wolfgang H, Öfner D. Cumulative Incidence of Permanent Stoma After Sphincter Preserving Low Anterior Resection of Mid and Low Rectal Cancer. Diseases of the Colon & Rectum. 2013;56(10):1134-42.
- [Background] Jørgensen JB, Erichsen R, Pedersen BG, Laurberg S, Iversen LH. Stoma reversal after intended restorative rectal cancer resection in Denmark: nationwide population-based study. BJS Open. 2020;4(6):1162-71.
- [Background] Xu X, Zhong H, You J, Ren M, Fingerhut A, Zheng M, et al. Revolutionizing sphincter preservation in ultra-low rectal cancer: exploring the potential of transanal endoscopic intersphincteric resection (taE-ISR): a propensity score-matched cohort study. Int J Surg. 2024;110(2):709-20.
- [Background] Back E, Häggström J, Holmgren K, Haapamäki MM, Matthiessen P, Rutegård J, et al. Permanent stoma rates after anterior resection for rectal cancer: risk prediction scoring using preoperative variables. Br J Surg. 2021;108(11):1388-95.
- [Background] Gadan S, Floodeen H, Lindgren R, Rutegård M, Matthiessen P. What is the risk of permanent stoma beyond 5 years after low anterior resection for rectal cancer? A 15-year follow-up of a randomized trial. Colorectal Dis. 2020;22(12):2098-104.
- [Background] Biondo S, Barrios O, Trenti L, Espin E, Bianco F, Falato A, et al. Long-Term Results of 2-Stage Turnbull-Cutait Pull-Through Coloanal Anastomosis for Low Rectal Cancer: A Randomized Clinical Trial. JAMA Surg. 2024;159(9):990-6.
- [Background] Biondo S, Trenti L, Espin E, Bianco F, Barrios O, Falato A, et al. Two-Stage Turnbull-Cutait Pull-Through Coloanal Anastomosis for Low Rectal Cancer: A Randomized Clinical Trial. JAMA Surg. 2020;155(8):e201625.
- [Background] La Raja C, Foppa C, Maroli A, Kontovounisios C, Ben David N, Carvello M, et al. Surgical outcomes of Turnbull-Cutait delayed coloanal anastomosis with pull-through versus immediate coloanal anastomosis with diverting stoma after total mesorectal excision for low rectal cancer: a systematic review and meta-analysis. Tech Coloproctol. 2022;26(8):603-13.
- [Background] Beirens K, Penninckx F. Defunctioning stoma and anastomotic leak rate after total mesorectal excision with coloanal anastomosis in the context of PROCARE. Acta Chir Belg. 2012;112(1):10-4.
- [Background] Guo Y, He L, Tong W, Ren S, Chi Z, Tan K, et al. Intersphincteric resection following robotic-assisted versus laparoscopy-assisted total mesorectal excision for middle and low rectal cancer: a multicentre propensity score analysis of 1571 patients. Int J Surg. 2024;110(4):1904-12.
- [Background] Schiessel R, Karner-Hanusch J, Herbst F, Teleky B, Wunderlich M. Intersphincteric resection for low rectal tumours. Br J Surg. 1994;81(9):1376-8.
- [Background] Rullier E, Denost Q, Vendrely V, Rullier A, Laurent C. Low rectal cancer: classification and standardization of surgery. Dis Colon Rectum. 2013;56(5):560-7.
- [Background] Parks AG. Transanal technique in low rectal anastomosis. Proc R Soc Med. 1972;65(11):975-6.
- [Background] Cutait DE, Figliolini FJ. A new method of colorectal anastomosis in abdominoperineal resection. Diseases of the Colon & Rectum. 1961;4(5):335-42.
- [Background] Turnbull RB, Cuthbertson A. Abdominorectal Pull-Through Resection for Cancer and for Hirschsprung's Disease. Delayed Posterior Colorectal Anastomosis. 1961;28(2):109-15.